# Double-blind randomized controlled study of linoleic acid supplementation for 1 year in patients with cystic fibrosis.

### -Influence on clinical status and metabolism.

## -NETwork study of LA supplementation in CF patients (NETLACF)

The study is registered at ClinTrial.gov ID #NCT04531410

**Funding:** European Society of Pediatric Gastroenterology and Nutrition; Swedish CF Association; Heart-Lung Foundation; Erica Lederhausen's Foundation.

The supplement was generously provided by AAK Ltd, Karlshamn/Copenhagen, Sweden/Denmark.

Updated 20241110

### admincontrol

2020-02871.pdf

Signers:

Name

Methods

Date

RIKARD BAKELIN

BANKID

2020-06-17 10.36 GMT+2

This document package contains: -

Front page (this page) -

The original document(s) -

The electronic signatures. These are not visible in the document,

but are electronically integrated.

We hereby certify that the English
translation corresponds to the Swedish
original document:

Amica April Patricia Degnell
Monica Ahlberg
08-524 81007

08-524 81007

Dnr 2020-02871

Stockholm division 2 medicine

#### **DECISION**

2020-06-16

#### **Applying Research Leader**

Karolinska Institutet

#### Researcher responsible for the project

Karl Ekwall

#### **Project title**

Double-blind controlled randomised study of fatty acid supplementation in cystic fibrosis and its influence on clinical status and metabolism.

#### Present change

Application registered 2020-05-26. Basic application approved 2019-01-16 by the Stockholm division 2 medicine with reference number 2019-00359.

The Ethical Appeal Board decides according to the decision below.

#### **Decision**

The Ethical Appeal Board approves the research which is described in the application for change.

On behalf of the Ethical Appeal Board

Rikard Backelin,

Chairman

The decision has been made after presentation of the report by the scientific secretary Gabriela Spulber.

#### The decision is sent to

Responsible researcher: Birgitta Strandvik

The Ethical Appeal Board

registrator@etikprovning.se / 010 4750800 / Box 2110, 75002 Uppsala / etikprovning.se